CLINICAL TRIAL: NCT05950737
Title: Sentinel Node Biopsy in Early Oral Cancers a Tertiary Cancer Centre Experience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Richa Vaish, Professor, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4205
Record Dates: First submitted 2023-07-07; First posted 2023-07-18 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Oral Cavity Squamous Cell Carcinoma
Keywords: oral neoplasm; sentinel node biopsy; node negative
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- sentinel node biopsy (Experimental): All patients have undergone completion neck dissection following SNB in the process of standardization. The SNB was localized by peritumoral infiltration of the nano colloid, followed by dynamic planar imaging for 30 minutes, and then SPECT was performed. The surgery was performed on the same day within 6 hours of localisation, and intraoperatively, either methylene blue or indocyanine green was used as an adjunct. Appropriately labelled sentinel nodes were assessed on the frozen section, which was then sectioned into 2-3mm slices perpendicular to the longest axis of the node and submitted entirely for microscopic evaluation. A minimum of 2 sections were evaluated, one stained with Toluidine blue and the other with rapid Haematoxylin and Eosin (HE) stain. The nodes were subsequently subjected to histopathological processing.
  Interventions: Procedure: Sentinel node biopsy

INTERVENTIONS:
Procedure: Sentinel node biopsy — All patients have undergone completion neck dissection following SNB in the process of standardization.

SUMMARY:
Sentinel node biopsy is a suitable alternative to END and is recommended in standard guidelines. Investigators have been doing SNB in their department to standardize the process for the last two years. This study aims to analyze the diagnostic accuracy of the SNB performed to standardize the procedure at their institute.

DETAILED DESCRIPTION:
Elective neck dissection (END) is the standard of care in node-negative early oral cancers.

However, it is associated with morbidity predominantly of shoulder dysfunction. Moreover, nearly 55-70% are true node-negative and are over-treated with this approach. Attempts have been made to overcome this limitation and to identify true node-negative patients. Sentinel node biopsy has shown the highest diagnostic accuracy among all other options. The SN is the first echelon node that drains directly through the lymphatics from the primary tumour. The principle of SNB is based on the fact that since it is the first echelon node, it would be the first site of regional metastasis. Therefore, the metastasis is unlikely to involve other nodal levels if the SNB is negative. It is the standard of care in breast cancers and melanoma. The concept made its way into oral cavity tumours and has been explored for over a decade in this setting. The results of the multi-institutional trial by Civantos et al. reported a high NPV of 94% of this procedure in early oral cancers that were node negative. Since then, various meta-analyses have shown that SNB has a high NPV making it a strong diagnostic modality. Schilling et al. reported the 3-year results of SNB in oral cancers in a multicentric study comprising 415 patients. The authors successfully identified the SN in 99.5% of cases and reported an FNR of 14%, which was high. Despite this, the study showed a high 3-year-disease-specific survival of 94%. Recently published Phase III Randomized controlled trials have shown that the overall survival of sentinel node biopsy is comparable to END with lesser morbidity in shoulder dysfunction. The advantage of the procedure is that only 25-30% of the patients who are SNB positive need to undergo neck dissection, and it spares unnecessary neck clearance and hence limits the morbidity in the remaining 70-75% of cases. SNB is a suitable alternative to END and is recommended in standard guidelines. However, SNB has a learning curve, it is recommended that the process be standardized, and the team should perform adequate SNB, followed by the completion of neck dissection before sparing the neck based on SNB. Investigators have been doing SNB in their department to standardize the process following the publication of level I evidence. This study aims to analyze the diagnostic accuracy of the SNB performed to standardize the procedure at the investigator's institute.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years of age,
2. Biopsy-proven invasive squamous cell carcinoma involving site among tongue and buccal mucosa
3. T1 and T2 lesions as per AJCC TNM classification
4. Clinicoradiologically node negative
5. Amenable to per oral excision

Exclusion Criteria:

1. Upper alveolar or palatal lesions
2. Large heterogeneous leukoplakia or other premalignant lesion
3. T3/T4 lesions
4. Lesions requiring raising of cheek flap to access for excision

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the SNB | Through study completion, an average of 2 year
  Sensitivity, specificity, negative predictive value, positive predictive value, False negative rate, SNB identification rate

SECONDARY OUTCOMES:
To study the pattern of metastasis in sentinel and non-sentinel nodes | Through study completion, an average of 2 year
  Level-wise frequency of SN metastasis, Frequency of metastasis in the SN basin, Frequency of metastasis to extra sentinel nodal basin

CONTACTS AND LOCATIONS:
Overall Officials: Richa Vaish, MS. M.Ch, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vaish R, Hawaldar R, Gupta S, Dandekar M, Shah S, Chaukar D, Pantvaidya G, Deshmukh A, Chaturvedi P, Pai P, Nair D, Nair S, Thakur M, Ghosh-Laskar S, Agarwal JP, D'Cruz AK. N0 neck trial: Does intensification of follow-up (Ultrasound + Physical Examination) influence outcomes in early-stage oral cancer? Eur J Cancer. 2024 Jun;204:114064. doi: 10.1016/j.ejca.2024.114064. Epub 2024 Apr 16. PMID 38705028
- [Background] D'Cruz AK, Vaish R, Kapre N, Dandekar M, Gupta S, Hawaldar R, Agarwal JP, Pantvaidya G, Chaukar D, Deshmukh A, Kane S, Arya S, Ghosh-Laskar S, Chaturvedi P, Pai P, Nair S, Nair D, Badwe R; Head and Neck Disease Management Group. Elective versus Therapeutic Neck Dissection in Node-Negative Oral Cancer. N Engl J Med. 2015 Aug 6;373(6):521-9. doi: 10.1056/NEJMoa1506007. Epub 2015 May 31. PMID 26027881
- [Background] Civantos FJ, Zitsch RP, Schuller DE, Agrawal A, Smith RB, Nason R, Petruzelli G, Gourin CG, Wong RJ, Ferris RL, El Naggar A, Ridge JA, Paniello RC, Owzar K, McCall L, Chepeha DB, Yarbrough WG, Myers JN. Sentinel lymph node biopsy accurately stages the regional lymph nodes for T1-T2 oral squamous cell carcinomas: results of a prospective multi-institutional trial. J Clin Oncol. 2010 Mar 10;28(8):1395-400. doi: 10.1200/JCO.2008.20.8777. Epub 2010 Feb 8. PMID 20142602
- [Background] Thompson CF, St John MA, Lawson G, Grogan T, Elashoff D, Mendelsohn AH. Diagnostic value of sentinel lymph node biopsy in head and neck cancer: a meta-analysis. Eur Arch Otorhinolaryngol. 2013 Jul;270(7):2115-22. doi: 10.1007/s00405-012-2320-0. Epub 2012 Dec 22. PMID 23263205
- [Background] Mallo Magarinos M, Suarez Ajuria M, Marichalar Mendia X, Alvarez-Calderon Iglesias O, Chamorro Petronacci CM, Garcia Garcia A, Perez Sayans M. Diagnostic yield of sentinel lymph node biopsy in oral squamous cell carcinoma T1/T2-N0: systematic review and meta-analysis. Int J Oral Maxillofac Surg. 2021 Oct;50(10):1271-1279. doi: 10.1016/j.ijom.2021.01.020. Epub 2021 Feb 16. PMID 33602650
- [Background] Yang Y, Zhou J, Wu H. Diagnostic value of sentinel lymph node biopsy for cT1/T2N0 tongue squamous cell carcinoma: a meta-analysis. Eur Arch Otorhinolaryngol. 2017 Nov;274(11):3843-3852. doi: 10.1007/s00405-017-4740-3. Epub 2017 Sep 12. PMID 28900723
- [Background] Schilling C, Stoeckli SJ, Haerle SK, Broglie MA, Huber GF, Sorensen JA, Bakholdt V, Krogdahl A, von Buchwald C, Bilde A, Sebbesen LR, Odell E, Gurney B, O'Doherty M, de Bree R, Bloemena E, Flach GB, Villarreal PM, Fresno Forcelledo MF, Junquera Gutierrez LM, Amezaga JA, Barbier L, Santamaria-Zuazua J, Moreira A, Jacome M, Vigili MG, Rahimi S, Tartaglione G, Lawson G, Nollevaux MC, Grandi C, Donner D, Bragantini E, Dequanter D, Lothaire P, Poli T, Silini EM, Sesenna E, Dolivet G, Mastronicola R, Leroux A, Sassoon I, Sloan P, McGurk M. Sentinel European Node Trial (SENT): 3-year results of sentinel node biopsy in oral cancer. Eur J Cancer. 2015 Dec;51(18):2777-84. doi: 10.1016/j.ejca.2015.08.023. Epub 2015 Nov 18. PMID 26597442
- [Background] Garrel R, Poissonnet G, Moya Plana A, Fakhry N, Dolivet G, Lallemant B, Sarini J, Vergez S, Guelfucci B, Choussy O, Bastit V, Richard F, Costes V, Landais P, Perriard F, Daures JP, de Verbizier D, Favier V, de Boutray M. Equivalence Randomized Trial to Compare Treatment on the Basis of Sentinel Node Biopsy Versus Neck Node Dissection in Operable T1-T2N0 Oral and Oropharyngeal Cancer. J Clin Oncol. 2020 Dec 1;38(34):4010-4018. doi: 10.1200/JCO.20.01661. Epub 2020 Oct 14. PMID 33052754
- [Background] Hasegawa Y, Tsukahara K, Yoshimoto S, Miura K, Yokoyama J, Hirano S, Uemura H, Sugasawa M, Yoshizaki T, Homma A, Chikamatsu K, Suzuki M, Shiotani A, Matsuzuka T, Kohno N, Miyazaki M, Oze I, Matsuo K, Kosuda S, Yatabe Y; HNCMM Research Group. Neck Dissections Based on Sentinel Lymph Node Navigation Versus Elective Neck Dissections in Early Oral Cancers: A Randomized, Multicenter, and Noninferiority Trial. J Clin Oncol. 2021 Jun 20;39(18):2025-2036. doi: 10.1200/JCO.20.03637. Epub 2021 Apr 20. PMID 33877855
- [Background] Vaish R, Mittal N, Mahajan A, Rane SU, Agrawal A, D'Cruz AK. Sentinel node biopsy in node negative early oral cancers: Solution to the conundrum! Oral Oncol. 2022 Nov;134:106070. doi: 10.1016/j.oraloncology.2022.106070. Epub 2022 Aug 18. PMID 35988294
- [Background] Vaish R. Shifting Paradigm of the Management of Node-Negative Neck in Early Oral Cancers: Where do we Stand Today? Indian J Med Paediatr Oncol 2022; 43(01): 092-094 DOI: 10.1055/s-0042-1742637